CLINICAL TRIAL: NCT04079790
Title: A Phase I, Double-Blind, Two-Part, Sequential Study to Evaluate the Pharmacokinetics of Gepotidacin Tablets in Healthy Adult and Adolescent Participants
Brief Title: Pharmacokinetics of Gepotidacin Tablets in Adults and Adolescents Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 209611
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Infections, Bacterial
Keywords: GSK2140944; Gepotidacin; Pharmacokinetics; Healthy Adult; Healthy adolescent
MeSH Terms: conditions — Bacterial Infections | interventions — gepotidacin

STUDY DESIGN:
Intervention Model Description: Part 1 is a 3-period, fixed-sequence study of a single 1500-mg dose (Period 1) and two 3000-mg doses of gepotidacin at Hours 0 and 12 (Period 2) and Hours 0 and 6 (Period 3) in healthy adult subjects. Part 2 is a 2-period, fixed sequence study of a single 1500 mg dose (Period 1) of gepotidacin and two 3000 mg doses (Period 2) of gepotidacin in healthy adolescent subjects. .
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects receiving Gepotidacin in Part 1 (Experimental): Healthy adult subjects will receive a single oral dose of gepotidacin 1500 mg (2 X 750 mg, treatment A), tablets, on Day 1 of Period 1; two oral doses of gepotidacin 3000 mg (4 x 750 mg, Treatment C), tablets, at 0 and 12 hours on Day 5 of Period 2; and two oral doses of gepotidacin 3000 mg (4 x 750 mg, treatment E), tablets, at 0 and 6 hours on Day 9 of Period 3.
  Interventions: Drug: Gepotidacin
- Subjects receiving Placebo in Part 1 (Placebo Comparator): Healthy adult subjects will receive a single oral dose of matching placebo (treatment B), tablets, on Day 1 of Period 1; two oral doses of matching placebo (treatment D), tablets, at 0 and 12 hours on Day 5 of Period 2; and two oral doses of matching placebo (treatment F), tablets, at 0 and 6 hours on Day 9 of Period 3.
  Interventions: Drug: Placebo
- Subjects receiving Gepotidacin in Part 2 (Experimental): Healthy adolescent subjects will receive a single oral dose of gepotidacin 1500 mg (2 x 750 mg, treatment A), tablets, on Day 1 of Period 1; and two oral doses of gepotidacin 3000 mg (4 x 750 mg, treatment G), tablets, at 0 and 6 hours on Day 1 of Period 2.
  Interventions: Drug: Gepotidacin
- Subjects receiving Placebo in Part 2 (Placebo Comparator): Healthy adolescent subjects will receive a single oral dose of matching placebo (treatment B), tablets on Day 1 of Period 1; and two oral doses of matching placebo (treatment H), tablets at 0 and 6 hours on Day 1 of Period 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gepotidacin — Tablets containing gepotidacin mesylate with a unit dose of 750 mg will be administered orally with 240 milliliter (mL) of water.
  Arms: Subjects receiving Gepotidacin in Part 1; Subjects receiving Gepotidacin in Part 2
Drug: Placebo — Tablets containing unit dose of placebo matching of gepotidacin will be administered orally with 240 mL of water.
  Arms: Subjects receiving Placebo in Part 1; Subjects receiving Placebo in Part 2

SUMMARY:
This is double-blind, randomized, sequential, two part study. Part 1 is a 3 periods, fixed-sequence study and will be conducted to evaluate the pharmacokinetics, safety, and tolerability of the gepotidacin tablet in healthy adult subjects. Part 2 is a 2 periods, fixed-sequence study and will evaluate the pharmacokinetics, safety, and tolerability of the gepotidacin tablet in healthy adolescent subjects. The primary purpose of Part 1 is to evaluate the pharmacokinetics of a single 1500 milligram (mg) dose and two 3000 mg doses of gepotidacin given 6 and 12 hours apart in adult subjects; Part 2 is to evaluate the pharmacokinetics of a single 1500 mg dose and two 3000 mg doses of gepotidacin given at a dosing interval (to be determined based on the pharmacokinetic and safety results from Part 1) in adolescent subjects. The duration of Part A will be approximately 47 days and 52 days for Part 2.

ELIGIBILITY:
Inclusion Criteria

* Subjects in Part 1 must be >=18 to <=64 years of age inclusive, at the time of signing the informed consent.
* Subjects in Part 2 must be >=12 to <18 years of age inclusive, at the time of signing the informed consent/assent.
* Subjects who are healthy as determined by the investigator or medically qualified designee based on medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead ECG results <450 millisecond (msec). A subject with clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the investigator feels and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=40 kilogram (kg) and body mass index (BMI) within the range 18.5 - 32.0 kg per square meter (inclusive).
* Male and/or female.
* Female subjects: A female subject is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: a) Is not a woman of childbearing potential (WOCBP), or b) Is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of <1% for at least 30 days prior to dosing until completion of the follow-up visit. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. A WOCBP must have a highly sensitive negative pregnancy test before the first dose of study intervention.
* Capable of giving signed informed consent/assent which includes compliance with the requirements and restrictions listed in the informed consent form/assent and protocol.

Exclusion Criteria

* Clinically significant abnormality in the past medical history or at the screening physical examination that in the investigator's opinion may place the subject at risk or interfere with outcome variables of the study. This includes, but is not limited to, history or current cardiac, hepatic, renal, neurologic, gastrointestinal (GI), respiratory, hematologic, or immunologic disease.
* Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention, or any other condition that may place the subject at risk, in the opinion of the investigator.
* Female subject has a positive pregnancy test result or is lactating at screening or upon admission to the clinic.
* Use of any systemic antibiotic within 30 days of screening.
* Within 2 months before screening, either a confirmed history of Clostridium difficile diarrhea infection or a past positive of Clostridium difficile toxin test.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of drug and/or alcohol abuse within 6 months before screening, as determined by the investigator, or has a positive drug screen at screening or upon admission to the clinic.
* History of sensitivity to any of the study drug, components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline medical monitor contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinic uses heparin to maintain intravenous cannula patency).
* Subject must abstain from taking prescription or non-prescription drugs (except for hormonal contraceptives and/or acetaminophen), vitamins, and dietary or herbal supplements, within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to study intervention until completion of the follow-up visit, unless, in the opinion of the investigator and sponsor, the medication will not interfere with the study. Any exceptions will be discussed with the sponsor or medical monitor on a case-by-case basis and the reasons will be documented.
* Previous exposure to gepotidacin within 12 months prior to starting study intervention.
* Subject has participated in a clinical trial and has received an investigational product prior to gepotidacin administration within 30 days, 5 half-lives, or twice the duration of the biological effect of investigational product (whichever is longer).
* Presence of hepatitis B surface antigen or positive hepatitis C antibody test result at screening or within 3 months prior to starting study intervention.
* ALT >1.5 * upper limit of normal (ULN).
* Bilirubin >1.5 * ULN (isolated bilirubin >1.5 * ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* History of any kidney disease or current or chronic history of impaired renal function as indicated by an estimated creatinine clearance <60 milliliter per minute (mL/min).
* A positive test for human immunodeficiency virus antibody.
* History of regular alcohol consumption within 6 months of screening defined as an average weekly intake of >21 units (or an average daily intake of >3 units) for males or an average weekly intake of >14 units (or an average daily intake >2 units) for females. One unit is equivalent to 270 mL of full strength beer, 470 mL of light beer, 30 mL of spirits, or 100 mL of wine.
* Urinary cotinine level indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 3 months before screening.
* Clinically significant abnormal findings in serum chemistry, hematology, or urinalysis results obtained at screening or Day -1.
* Baseline corrected QT interval using the Fridericia formula (QTcF) of >450 msec.
* Subject has donated blood in excess of 500 mL within 12 weeks prior to dosing or participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56-day period.
* Subject is unable to comply with all study procedures, in the opinion of the investigator.
* Subject should not participate in the study, in the opinion of the investigator or sponsor.

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Barth A, Hossain M, Brimhall DB, Perry CR, Tiffany CA, Xu S, Dumont EF. Pharmacokinetics of Oral Formulations of Gepotidacin (GSK2140944), a Triazaacenaphthylene Bacterial Type II Topoisomerase Inhibitor, in Healthy Adult and Adolescent Participants. Antimicrob Agents Chemother. 2022 Jan 18;66(1):e0126321. doi: 10.1128/AAC.01263-21. Epub 2021 Oct 11. PMID 34633853

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-part, double-blind, randomized, sequential study to evaluate pharmacokinetics of Gepotidacin in healthy adult and adolescent participants. The study was conducted at a single center in the United States.
Pre-assignment Details: A total of 34 participants were randomized in this study (Randomized Population): 16 adult participants in Part 1 and 18 adolescent participants in Part 2.
Groups:
- Gepotidacin (A/C/E): Adult participants were randomized to receive a single dose of gepotidacin 1500 milligrams (mg) (Treatment A) on Day 1 of Period 1 followed by two doses of gepotidacin 3000 mg separated by 12 hours (Treatment C) on Day 5 of Period 2, and two doses of gepotidacin 3000 mg separated by 6 hours (Treatment E) on Day 9 of Period 3. All doses were administered orally with water after consumption of food.
- Placebo (B/D/F): Adult participants were randomized to receive a single dose of gepotidacin matching placebo (Treatment B) on Day 1 of Period 1 followed by two doses of gepotidacin matching placebo separated by 12 hours (Treatment D) on Day 5 of Period 2, and two doses of gepotidacin matching placebo separated by 6 hours (Treatment F) on Day 9 of Period 3. All doses were administered orally with water after consumption of food.
- Gepotidacin (A/G): Adolescent participants were randomized to receive a single dose of gepotidacin 1500 mg (Treatment A) on Day 1 of Period 1 followed by two doses of gepotidacin 3000 mg separated by 6 hours (Treatment G) on Day 1 of Period 2. All doses were administered orally with water after consumption of food.
- Placebo (B/H): Adolescent participants were randomized to receive a single dose of gepotidacin matching placebo (Treatment B) on Day 1 of Period 1 followed by two doses of gepotidacin matching placebo separated by 6 hours (Treatment H) on Day 1 of Period 2. All doses were administered orally with water after consumption of food.
Period: Part 1, Period 1(Day 1 to Day 4)
Arm/Group | Gepotidacin (A/C/E) | Placebo (B/D/F) | Gepotidacin (A/G) | Placebo (B/H)
Started | 14 | 2 | 0 | 0
Completed | 13 | 2 | 0 | 0
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Period: Part 1, Period 2 (Day 5 to Day 8)
Arm/Group | Gepotidacin (A/C/E) | Placebo (B/D/F) | Gepotidacin (A/G) | Placebo (B/H)
Started | 13 | 2 | 0 | 0
Completed | 13 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 1, Period 3 (Day 9 to Day 11)
Arm/Group | Gepotidacin (A/C/E) | Placebo (B/D/F) | Gepotidacin (A/G) | Placebo (B/H)
Started | 13 | 2 | 0 | 0
Completed | 13 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Part 2, Period 1 (Day 1 to Day 3)
Arm/Group | Gepotidacin (A/C/E) | Placebo (B/D/F) | Gepotidacin (A/G) | Placebo (B/H)
Started | 0 | 0 | 15 | 3
Completed | 0 | 0 | 12 | 3
Not Completed | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Unable to swallow | 0 | 0 | 2 | 0
Period: Part 2, Period 2 (Day 1 to Day 3)
Arm/Group | Gepotidacin (A/C/E) | Placebo (B/D/F) | Gepotidacin (A/G) | Placebo (B/H)
Started | 0 | 0 | 12 | 3
Completed | 0 | 0 | 12 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gepotidacin (A/C/E) | Placebo (B/D/F) | Gepotidacin (A/G) | Placebo (B/H) | Total
Number analyzed (Participants) | 14 | 2 | 14 | 3 | 33
Age, Categorical [Count of Participants; unit: Participants] — Baseline characteristics is presented for Safety Population which consisted of all participants who took at least 1 dose of study intervention. This population was used for demographic and safety summaries. One participant was randomized to Gepotidacin (A/G) arm but was unable to swallow the tablet and was not a part of Safety Population.
  Participants
    <=18 years | 0 | 0 | 14 | 3 | 17
    Between 18 and 65 years | 14 | 2 | 0 | 0 | 16
    >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population: One participant was randomized to Gepotidacin (A/G) arm but was unable to swallow the tablet and was not a part of safety population
  Participants
    Female | 6 | 1 | 4 | 1 | 12
    Male | 8 | 1 | 10 | 2 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Safety Population: One participant was randomized to Gepotidacin (A/G) arm but was unable to swallow the tablet and was not a part of safety population.
  Participants
    Asian- Central/South Asian Heritage | 1 | 0 | 1 | 0 | 2
    Black or African American | 6 | 0 | 6 | 1 | 13
    White-Arabic/North African Heritage | 1 | 0 | 0 | 0 | 1
    White-White/Caucasian/European Heritage | 6 | 2 | 5 | 2 | 15
    Multiple | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1- Period 1: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to Time of the Last Quantifiable Concentration (AUC[0-t]) After Single Dose Administration of Gepotidacin 1500 mg
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of gepotidacin. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter Population consisted of all participants in the PK Population (participants who received at least 1 dose of gepotidacin and had evaluable post-dose plasma concentration data for gepotidacin), for whom valid and evaluable PK parameters were derived.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 1: Gepotidacin 1500 mg: Adult participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours*micrograms per milliliter | 19.69 (17.6)

2. Primary Outcome: Part 1- Period 1: Area Under the Concentration-time Curve From Time 0 (Pre-dose) Extrapolated to Infinite Time (AUC[0-infinity]) After Single Dose Administration of Gepotidacin 1500 mg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours*micrograms per milliliter | 20.15 (16.8)

3. Primary Outcome: Part 1- Period 1: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to 24 Hours Post-dose (AUC[0-24]) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours*micrograms per milliliter | 18.66 (19.5)

4. Primary Outcome: Part 1- Period 1: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to 48 Hours Post-dose (AUC[0-48]) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours*micrograms per milliliter | 19.72 (17.6)

5. Primary Outcome: Part 1- Period 1: Maximum Observed Concentration (Cmax) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Micrograms per milliliter | 3.574 (38.1)

6. Primary Outcome: Part 1- Period 2: AUC(0-t) Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 1: Gepotidacin 3000 mg 12 Hour Interval: Participants were administered two doses of gepotidacin 3000 mg separated by 12 hours (Dose 1 at Hour 0 and dose 2 at Hour 12)
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 91.21 (22.6)

7. Primary Outcome: Part 1- Period 3: AUC(0-t) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 1: Gepotidacin 3000 mg 6 Hour Interval: Participants were administered two doses of gepotidacin 3000 mg separated by 6 hours (Dose 1 at Hour 0 and dose 2 at Hour 6)
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 87.09 (26.3)

8. Primary Outcome: Part 1- Period 2: Area Under the Concentration-time Curve From Time 0 (Pre-dose) to Time Tau (Tau=12) (AUC[0-tau]) Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8 and 12 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter
  Dose 1 | 38.15 (24.3)
  Dose 2 | 44.41 (22.8)

9. Primary Outcome: Part 1- Period 3: AUC(0-tau) (Tau=6) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4 and 6 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter
  Dose 1 | 24.09 (33.6)
  Dose 2 | 40.13 (29.5)

10. Primary Outcome: Part 1- Period 2: AUC(0-24) Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20 and 24 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 83.45 (22.7)

11. Primary Outcome: Part 1- Period 3: AUC(0-24) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18 and 24 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 82.43 (27.3)

12. Primary Outcome: Part 1- Period 2: AUC(0-48) Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 90.53 (22.7)

13. Primary Outcome: Part 1- Period 3: AUC(0-48) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 86.49 (26.4)

14. Primary Outcome: Part 1- Period 2: Accumulation Ratio for Cmax (RoCmax) Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio was calculated as Cmax after the second dose divided by Cmax after the first dose.
Time Frame: as for outcome 6
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Ratio | 1.109 (30.6)

15. Primary Outcome: Part 1- Period 2: Accumulation Ratio for AUC (RoAUC) Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio was calculated as AUC(0-tau) after the second dose, where 0 is the timepoint prior to second dose, divided by AUC(0-tau) after the first dose, where 0 is the predose timepoint prior to the first dose.
Time Frame: as for outcome 6
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Ratio | 1.164 (12.7)

16. Primary Outcome: Part 1- Period 3: RoCmax Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: as for outcome 14
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Ratio | 1.544 (25.9)

17. Primary Outcome: Part 1- Period 3: RoAUC Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: as for outcome 15
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Ratio | 1.666 (25.9)

18. Primary Outcome: Part 1- Period 2: Cmax Following Two Doses of Gepotidacin 3000 mg Administered at 12 Hour Dosing Interval
Description: as for outcome 2
Time Frame: as for outcome 6
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Micrograms per milliliter
  Dose 1 | 9.937 (24.2)
  Dose 2 | 11.02 (28.1)

19. Primary Outcome: Part 1- Period 3: Cmax Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Dosing Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Groups:
- Part1: Gepotidacin 3000 mg 6 Hour Interval: Participants were administered two doses of gepotidacin 3000 mg separated by 6 hours (Dose 1 at Hour 0 and dose 2 at Hour 6)
Arm/Group | Part1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Micrograms per milliliter
  Dose 1 | 8.423 (41.8)
  Dose 2 | 13.01 (28.6)

20. Primary Outcome: Part 2- Period 1: AUC(0-t) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 2: Gepotidacin 1500 mg: Adolescent participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 23.27 (21.6)

21. Primary Outcome: Part 2- Period 1: AUC(0-infinity) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 23.79 (20.9)

22. Primary Outcome: Part 2- Period 1: AUC(0-24) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 and 24 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 22.06 (22.6)

23. Primary Outcome: Part 2- Period 1: AUC(0-48) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 23.27 (21.6)

24. Primary Outcome: Part 2- Period 1: Cmax After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Micrograms per milliliter | 4.523 (29.5)

25. Primary Outcome: Part 2- Period 2: AUC(0-t) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 2-Gepotidacin 3000 mg 6 Hour Interval: Participants were administered two doses of gepotidacin 3000 mg separated by 6 hours (Dose 1 at Hour 0 and dose 2 at Hour 6)
Arm/Group | Part 2-Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter | 115.6 (23.8)

26. Primary Outcome: Part 2- Period 2: AUC(0-tau) (Tau=6) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4 and 6 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 2: Gepotidacin 3000 mg 6 Hour Interval: Participants were administered two doses of gepotidacin 3000 mg separated by 6 hours (Dose 1 at Hour 0 and dose 2 at Hour 6)
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter
  Dose 1 | 32.37 (22.0)
  Dose 2 | 53.85 (26.7)

27. Primary Outcome: Part 2- Period 2: AUC(0-24) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18 and 24 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter | 111.4 (23.8)

28. Primary Outcome: Part 2- Period 2: AUC(0-48) Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter | 115.6 (23.8)

29. Primary Outcome: Part 2- Period 2: Cmax Following Two Doses of Gepotidacin 3000 mg Administered at 6 Hour Interval
Description: as for outcome 2
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Micrograms per milliliter
  Dose 1 | 10.86 (26.8)
  Dose 2 | 14.29 (29.5)

30. Primary Outcome: Part 1: Number of Participants With Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with common (>=5%) non-serious AEs and SAEs is presented.
Time Frame: Up to Day 19
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Placebo: Adult participants received a single oral dose of gepotidacin matching placebo on Day 1 of Period 1
- Part 1: Gepotidacin 3000 mg 12 Hour Interval: Adult participants were administered two doses of gepotidacin 3000 mg separated by 12 hours (Dose 1 at Hour 0 and dose 2 at Hour 12)
- Part 1: Gepotidacin 3000 mg 6 Hour Interval: Adult participants were administered two doses of gepotidacin 3000 mg separated by 6 hours (Dose 1 at Hour 0 and dose 2 at Hour 6)
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 14 | 13 | 13
Participants
  Common non-serious AEs | 0 | 1 | 10 | 9
  SAEs | 0 | 0 | 0 | 0

31. Primary Outcome: Part 2: Number of Participants With Non-serious AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with common (>=5%) non-serious AEs and SAEs are presented.
Time Frame: Up to Day 21
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Placebo: Adolescent participants received a single oral dose of gepotidacin matching placebo on Day 1 of Period 1
- Part 2: Gepotidacin 3000 mg 6 Hour Interval: Adolescent participants were administered two doses of gepotidacin 3000 mg separated by 6 hours (Dose 1 at Hour 0 and dose 2 at Hour 6)
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 14 | 12
Participants
  Common non-serious AEs | 2 | 9 | 12
  SAEs | 0 | 0 | 0

32. Primary Outcome: Part 1: Number of Participants With Hematology Toxicities of Grade 3 or Higher
Description: Blood samples were collected for the analysis of following hematology parameters: platelet count, red blood cell (RBC) count, hemoglobin, hematocrit, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), white blood cell (WBC) count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. The hematology abnormalities were graded using the Division of Microbiology and Infectious Diseases toxicity grading where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4=Life-threatening. Number of participants with a grade 3 or higher toxicity for any of the hematology parameter is presented.
Time Frame: Up to Day 19
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 14 | 13 | 13
Participants | 0 | 0 | 0 | 0

33. Primary Outcome: Part 2: Number of Participants With Hematology Toxicities of Grade 3 or Higher
Description: Blood samples were collected for the analysis of following hematology parameters: platelet count, RBC count, hemoglobin, hematocrit, MCV, MCH, WBC count, neutrophils, lymphocytes, monocytes, eosinophils and basophils. The hematology abnormalities were graded using the Division of Microbiology and Infectious Diseases toxicity grading where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4=Life-threatening. Number of participants with a grade 3 or higher toxicity for any of the hematology parameter is presented.
Time Frame: Up to Day 21
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 14 | 12
Participants | 0 | 0 | 0

34. Primary Outcome: Part 1: Number of Participants With Clinical Chemistry Toxicities of Grade 3 or Higher
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: blood urea nitrogen (BUN), creatinine, glucose (fasting), potassium, sodium, magnesium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total and direct bilirubin, creatine phosphokinase, calcium, chloride, carbon dioxide, total protein and albumin. The clinical chemistry abnormalities were graded using the Division of Microbiology and Infectious Diseases toxicity grading where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4=Life-threatening. Number of participants with a grade 3 or higher toxicity for any of the clinical chemistry parameter is presented
Time Frame: Up to Day 19
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 14 | 13 | 13
Participants | 0 | 0 | 0 | 0

35. Primary Outcome: Part 2: Number of Participants With Clinical Chemistry Toxicities of Grade 3 or Higher
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: BUN, creatinine, glucose (fasting), potassium, sodium, magnesium, AST, ALT, alkaline phosphatase, total and direct bilirubin, creatine phosphokinase, calcium, chloride, carbon dioxide, total protein and albumin. The clinical chemistry abnormalities were graded using the Division of Microbiology and Infectious Diseases toxicity grading where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4=Life-threatening. Number of participants with a grade 3 or higher toxicity for any of the clinical chemistry parameter is presented
Time Frame: Up to Day 21
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 14 | 12
Participants | 1 | 1 | 3

36. Primary Outcome: Part 1: Number of Participants With Urinalysis Toxicities of Grade 3 or Higher
Description: Urine samples were collected for the analysis of urine parameters including specific gravity, potential of hydrogen (pH), glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase. Toxicities were graded using the Division of Microbiology and Infectious Diseases toxicity grading where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4=Life-threatening. Number of participants with a grade 3 or higher toxicity for any of the urine parameter is presented
Time Frame: Up to Day 19
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 14 | 13 | 13
Participants | 0 | 0 | 0 | 0

37. Primary Outcome: Part 2: Number of Participants With Urinalysis Toxicities of Grade 3 or Higher
Description: Urine samples were collected for the analysis of urine parameters including specific gravity, pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase. Toxicities were graded using the Division of Microbiology and Infectious Diseases toxicity grading where Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe and Grade 4=Life-threatening. Number of participants with a grade 3 or higher toxicity for any of the urine parameter is presented
Time Frame: Up to Day 21
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 14 | 12
Participants | 0 | 0 | 0

38. Primary Outcome: Part 1: Number of Participants With Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) of Potential Clinical Importance
Description: SBP and DBP were measured in a semi-supine position after 5 minutes of rest. The potential clinically important range for vital signs were: SBP (lower: <85 and upper: >160 millimeters of mercury [mmHg]) and DBP (lower: <45 and upper: >100 mmHg).
Time Frame: Up to Day 19
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 14 | 13 | 13
Participants | 0 | 0 | 1 | 1

39. Primary Outcome: Part 2: Number of Participants With SBP and DBP of Potential Clinical Importance
Description: SBP and DBP were measured in a semi-supine position after 5 minutes of rest. The potential clinically important range for vital signs were: SBP (lower: <85 and upper: >160 mmHg) and DBP (lower: <45 and upper: >100 mmHg).
Time Frame: Up to Day 21
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 14 | 12
Participants | 0 | 0 | 0

40. Primary Outcome: Part 1: Number of Participants With Abnormal Heart Rate of Potential Clinical Importance
Description: Heart rate was measured in a semi-supine position after 5 minutes of rest. The potential clinically important range for heart rate was (lower:<40 and upper: >110 beats per minute).
Time Frame: Up to Day 19
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 14 | 13 | 13
Participants | 0 | 0 | 0 | 1

41. Primary Outcome: Part 2: Number of Participants With Abnormal Heart Rate of Potential Clinical Importance
Description: as for outcome 40
Time Frame: Up to Day 21
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 14 | 12
Participants | 0 | 1 | 0

42. Primary Outcome: Part 1: Period 1: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes. Twelve lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and corrected QT (QTc) intervals and calculated heart rate. Data for abnormal not clinically significant (NCS) and clinically significant (CS) ECG findings are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Predose, predose 2, predose 3, 0.5. 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12 hours on Day 1, 24, 36 hours on Day 2 and 48 hours on Day 3.
Population: Safety population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 2 | 14
Participants
  Abnormal, NCS, Day 1- predose, n= 2, 14 | 1 | 8
  Abnormal, CS, Day 1- predose, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- predose 2, n= 2, 14 | 1 | 11
  Abnormal, CS, Day 1-predose 2, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- predose 3, n= 2, 14 | 1 | 12
  Abnormal, CS, Day 1- predose 3, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 0.5 hours, n= 2, 14 | 0 | 7
  Abnormal, CS, Day 1- 0.5 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 1 hour, n= 2, 14 | 0 | 7
  Abnormal, CS, Day 1- 1 hour, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 1.5 hours, n= 2, 14 | 0 | 9
  Abnormal, CS, Day 1- 1.5 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 2 hours, n= 2, 14 | 0 | 9
  Abnormal, CS, Day 1- 2 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 2.5 hours, n= 2, 14 | 1 | 10
  Abnormal, CS, Day 1- 2.5 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 3 hours, n= 2, 14 | 0 | 8
  Abnormal, CS, Day 1- 3 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 4 hours, n= 2, 14 | 1 | 11
  Abnormal, CS, Day 1- 4 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 6 hours, n= 2, 14 | 1 | 9
  Abnormal, CS, Day 1- 6 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 8 hours, n= 2, 14 | 1 | 9
  Abnormal, CS, Day 1- 8 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 1- 12 hours, n= 2, 14 | 0 | 9
  Abnormal, CS, Day 1- 12 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 2- 24 hours, n= 2, 14 | 1 | 10
  Abnormal, CS, Day 2- 24 hours, n= 2, 14 | 0 | 0
  Abnormal, NCS, Day 2- 36 hours, n= 2, 13: number analyzed (Participants) | 2 | 13
  Abnormal, NCS, Day 2- 36 hours, n= 2, 13 | 0 | 5
  Abnormal, CS, Day 2- 36 hours, n= 2, 13: number analyzed (Participants) | 2 | 13
  Abnormal, CS, Day 2- 36 hours, n= 2, 13 | 0 | 0
  Abnormal, NCS, Day 3- 48 hours, n= 2, 13: number analyzed (Participants) | 2 | 13
  Abnormal, NCS, Day 3- 48 hours, n= 2, 13 | 1 | 11
  Abnormal, CS, Day 3- 48 hours, n= 2, 13: number analyzed (Participants) | 2 | 13
  Abnormal, CS, Day 3- 48 hours, n= 2, 13 | 0 | 0

43. Primary Outcome: Part 1: Period 2: Number of Participants With Abnormal 12-lead ECG Findings
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes. Twelve lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and QTc intervals and calculated heart rate. Data for abnormal NCS and CS ECG findings are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Predose, predose 2, predose 3, 0.5. 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 12.5, 13, 13.5, 14, 14.5, 15, 16, 18, 20 hours on Day 1, 24, 36 hours on Day 2, 48 and 60 hours on Day 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 2 | 13
Participants
  Abnormal, NCS, Day 1- predose | 2 | 8
  Abnormal, CS, Day 1- predose | 0 | 0
  Abnormal, NCS, Day 1- predose 2 | 2 | 8
  Abnormal, CS, Day 1-predose 2 | 0 | 0
  Abnormal, NCS, Day 1- predose 3 | 1 | 9
  Abnormal, CS, Day 1- predose 3 | 0 | 0
  Abnormal, NCS, Day 1- 0.5 hours | 1 | 9
  Abnormal, CS, Day 1- 0.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 1 hour | 1 | 10
  Abnormal, CS, Day 1- 1 hour | 0 | 0
  Abnormal, NCS, Day 1- 1.5 hours | 1 | 8
  Abnormal, CS, Day 1- 1.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 2 hours | 1 | 9
  Abnormal, CS, Day 1- 2 hours | 0 | 0
  Abnormal, NCS, Day 1- 2.5 hours | 1 | 7
  Abnormal, CS, Day 1- 2.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 3 hours | 1 | 9
  Abnormal, CS, Day 1- 3 hours | 0 | 0
  Abnormal, NCS, Day 1- 4 hours | 2 | 7
  Abnormal, CS, Day 1- 4 hours | 0 | 0
  Abnormal, NCS, Day 1- 6 hours | 1 | 9
  Abnormal, CS, Day 1- 6 hours | 0 | 0
  Abnormal, NCS, Day 1- 8 hours | 1 | 9
  Abnormal, CS, Day 1- 8 hours | 0 | 0
  Abnormal, NCS, Day 1- 12 hours | 1 | 8
  Abnormal, CS, Day 1- 12 hours | 0 | 0
  Abnormal, NCS, Day 1- 12.5 hours | 1 | 5
  Abnormal, CS, Day 1- 12.5 hours | 0 | 1
  Abnormal, NCS, Day 1- 13 hours | 1 | 8
  Abnormal, CS, Day 1- 13 hours | 0 | 0
  Abnormal, NCS, Day 1- 13.5 hours | 2 | 10
  Abnormal, CS, Day 1- 13.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 14 hours | 2 | 7
  Abnormal, CS, Day 1- 14 hours | 0 | 0
  Abnormal, NCS, Day 1- 14.5 hours | 2 | 9
  Abnormal, CS, Day 1- 14.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 15 hours | 1 | 8
  Abnormal, CS, Day 1- 15 hours | 0 | 0
  Abnormal, NCS, Day 1- 16 hours | 1 | 9
  Abnormal, CS, Day 1- 16 hours | 0 | 0
  Abnormal, NCS, Day 1- 18 hours | 1 | 11
  Abnormal, CS, Day 1- 18 hours | 0 | 0
  Abnormal, NCS, Day 1- 20 hours | 1 | 10
  Abnormal, CS, Day 1- 20 hours | 0 | 0
  Abnormal, NCS, Day 2- 24 hours | 1 | 9
  Abnormal, CS, Day 2- 24 hours | 0 | 0
  Abnormal, NCS, Day 2- 36 hours | 1 | 8
  Abnormal, CS, Day 2- 36 hours | 0 | 0
  Abnormal, NCS, Day 3- 48 hours | 1 | 11
  Abnormal, CS, Day 3- 48 hours | 0 | 0
  Abnormal, NCS, Day 3- 60 hours | 1 | 5
  Abnormal, CS, Day 3- 60 hours | 0 | 0

44. Primary Outcome: Part 1: Period 3: Number of Participants With Abnormal 12-lead ECG Findings
Description: as for outcome 43
Time Frame: Predose, predose 2, predose 3, 0.5. 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18 hours on Day 1, 24, 36 hours on Day 2, 48 and 60 hours on Day 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Placebo | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 2 | 13
Participants
  Abnormal, NCS, Day 1- predose | 1 | 11
  Abnormal, CS, Day 1- predose | 0 | 0
  Abnormal, NCS, Day 1- predose 2 | 0 | 9
  Abnormal, CS, Day 1-predose 2 | 0 | 0
  Abnormal, NCS, Day 1- predose 3 | 1 | 10
  Abnormal, CS, Day 1- predose 3 | 0 | 0
  Abnormal, NCS, Day 1- 0.5 hours | 1 | 9
  Abnormal, CS, Day 1- 0.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 1 hour | 1 | 9
  Abnormal, CS, Day 1- 1 hour | 0 | 0
  Abnormal, NCS, Day 1- 1.5 hours | 1 | 9
  Abnormal, CS, Day 1- 1.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 2 hours | 1 | 9
  Abnormal, CS, Day 1- 2 hours | 0 | 0
  Abnormal, NCS, Day 1- 2.5 hours | 0 | 8
  Abnormal, CS, Day 1- 2.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 3 hours | 1 | 9
  Abnormal, CS, Day 1- 3 hours | 0 | 0
  Abnormal, NCS, Day 1- 4 hours | 2 | 8
  Abnormal, CS, Day 1- 4 hours | 0 | 0
  Abnormal, NCS, Day 1- 6 hours | 2 | 7
  Abnormal, CS, Day 1- 6 hours | 0 | 0
  Abnormal, NCS, Day 1- 6.5 hours | 0 | 7
  Abnormal, CS, Day 1- 6.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 7 hours | 0 | 7
  Abnormal, CS, Day 1- 7 hours | 0 | 0
  Abnormal, NCS, Day 1- 7.5 hours | 0 | 10
  Abnormal, CS, Day 1- 7.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 8 hours | 1 | 11
  Abnormal, CS, Day 1- 8 hours | 0 | 0
  Abnormal, NCS, Day 1- 8.5 hours | 2 | 10
  Abnormal, CS, Day 1- 8.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 9 hours | 1 | 11
  Abnormal, CS, Day 1- 9 hours | 0 | 0
  Abnormal, NCS, Day 1- 10 hours | 2 | 8
  Abnormal, CS, Day 1- 10 hours | 0 | 0
  Abnormal, NCS, Day 1- 12 hours | 1 | 6
  Abnormal, CS, Day 1- 12 hours | 0 | 0
  Abnormal, NCS, Day 1- 14 hours | 0 | 7
  Abnormal, CS, Day 1- 14 hours | 0 | 0
  Abnormal, NCS, Day 1- 18 hours | 1 | 10
  Abnormal, CS, Day 1- 18 hours | 0 | 0
  Abnormal, NCS, Day 2- 24 hours | 1 | 8
  Abnormal, CS, Day 2- 24 hours | 0 | 0
  Abnormal, NCS, Day 2- 36 hours | 0 | 10
  Abnormal, CS, Day 2- 36 hours | 0 | 0
  Abnormal, NCS, Day 3- 48 hours | 1 | 10
  Abnormal, CS, Day 3- 48 hours | 0 | 0
  Abnormal, NCS, Day 3- 60 hours | 0 | 8
  Abnormal, CS, Day 3- 60 hours | 0 | 0

45. Primary Outcome: Part 2: Period 1: Number of Participants With Abnormal 12-lead ECG Findings
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes. Twelve lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and QTc intervals and calculated heart rate. Data for abnormal NCS and CS were presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 3 | 14
Participants
  Abnormal, NCS, Day 1- predose, n= 3, 14 | 1 | 4
  Abnormal, CS, Day 1- predose, n= 3, 14 | 0 | 0
  Abnormal, NCS, Day 1- predose 2, n= 3, 14 | 0 | 5
  Abnormal, CS, Day 1-predose 2, n= 3, 14 | 0 | 0
  Abnormal, NCS, Day 1- predose 3, n= 3, 14 | 0 | 4
  Abnormal, CS, Day 1- predose 3, n= 3, 14 | 0 | 0
  Abnormal, NCS, Day 1- 0.5 hours, n= 3, 14 | 0 | 5
  Abnormal, CS, Day 1- 0.5 hours, n= 3, 14 | 0 | 0
  Abnormal, NCS, Day 1- 1 hour, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 1 hour, n= 3, 13 | 0 | 7
  Abnormal, CS, Day 1- 1 hour, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 1 hour, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 1.5 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 1.5 hours, n= 3, 13 | 0 | 4
  Abnormal, CS, Day 1- 1.5 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 1.5 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 2 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 2 hours, n= 3, 13 | 0 | 4
  Abnormal, CS, Day 1- 2 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 2 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 2.5 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 2.5 hours, n= 3, 13 | 0 | 4
  Abnormal, CS, Day 1- 2.5 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 2.5 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 3 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 3 hours, n= 3, 13 | 1 | 6
  Abnormal, CS, Day 1- 3 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 3 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 4 hours, n= 3, 14 | 0 | 5
  Abnormal, CS, Day 1- 4 hours, n= 3, 14 | 0 | 0
  Abnormal, NCS, Day 1- 6 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 6 hours, n= 3, 13 | 0 | 6
  Abnormal, CS, Day 1- 6 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 6 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 8 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 8 hours, n= 3, 13 | 1 | 3
  Abnormal, CS, Day 1- 8 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 8 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 12 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 12 hours, n= 3, 13 | 0 | 6
  Abnormal, CS, Day 1- 12 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 12 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 24 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 24 hours, n= 3, 13 | 2 | 4
  Abnormal, CS, Day 1- 24 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 24 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 36 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 36 hours, n= 3, 13 | 0 | 3
  Abnormal, CS, Day 1- 36 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 36 hours, n= 3, 13 | 0 | 0
  Abnormal, NCS, Day 1- 48 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, NCS, Day 1- 48 hours, n= 3, 13 | 2 | 5
  Abnormal, CS, Day 1- 48 hours, n= 3, 13: number analyzed (Participants) | 3 | 13
  Abnormal, CS, Day 1- 48 hours, n= 3, 13 | 0 | 0

46. Primary Outcome: Part 2: Period 2: Number of Participants With Abnormal 12-lead ECG Findings
Description: A 12-lead ECG was recorded with the participant in a semi-supine position after a rest of at least 10 minutes. Twelve lead ECGs were obtained by using an automated ECG machine that measured PR, QRS, QT, and QTc intervals and calculated heart rate. Data for abnormal NCS and CS were presented CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: Predose, predose 2, predose 3, 0.5. 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18 hours on Day 1, 24, 36 hours on Day 2 and 48 hours on Day 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 3 | 12
Participants
  Abnormal, NCS, Day 1- predose | 1 | 6
  Abnormal, CS, Day 1- predose | 0 | 0
  Abnormal, NCS, Day 1- predose 2 | 1 | 7
  Abnormal, CS, Day 1-predose 2 | 0 | 0
  Abnormal, NCS, Day 1- predose 3 | 1 | 7
  Abnormal, CS, Day 1- predose 3 | 0 | 0
  Abnormal, NCS, Day 1- 0.5 hours | 1 | 6
  Abnormal, CS, Day 1- 0.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 1 hour | 1 | 6
  Abnormal, CS, Day 1- 1 hour | 0 | 0
  Abnormal, NCS, Day 1- 1.5 hours | 0 | 4
  Abnormal, CS, Day 1- 1.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 2 hours | 0 | 6
  Abnormal, CS, Day 1- 2 hours | 0 | 0
  Abnormal, NCS, Day 1- 2.5 hours | 0 | 5
  Abnormal, CS, Day 1- 2.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 3 hours | 0 | 5
  Abnormal, CS, Day 1- 3 hours | 0 | 0
  Abnormal, NCS, Day 1- 4 hours | 1 | 5
  Abnormal, CS, Day 1- 4 hours | 0 | 0
  Abnormal, NCS, Day 1- 6 hours | 1 | 3
  Abnormal, CS, Day 1- 6 hours | 0 | 0
  Abnormal, NCS, Day 1- 6.5 hours | 1 | 5
  Abnormal, CS, Day 1- 6.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 7 hours | 1 | 5
  Abnormal, CS, Day 1- 7 hours | 0 | 0
  Abnormal, NCS, Day 1- 7.5 hours | 0 | 3
  Abnormal, CS, Day 1- 7.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 8 hours | 0 | 3
  Abnormal, CS, Day 1- 8 hours | 0 | 0
  Abnormal, NCS, Day 1- 8.5 hours | 0 | 3
  Abnormal, CS, Day 1- 8.5 hours | 0 | 0
  Abnormal, NCS, Day 1- 9 hours | 0 | 4
  Abnormal, CS, Day 1- 9 hours | 0 | 0
  Abnormal, NCS, Day 1- 10 hours | 1 | 5
  Abnormal, CS, Day 1- 10 hours | 0 | 0
  Abnormal, NCS, Day 1- 12 hours | 0 | 4
  Abnormal, CS, Day 1- 12 hours | 0 | 0
  Abnormal, NCS, Day 1- 14 hours | 0 | 4
  Abnormal, CS, Day 1- 14 hours | 0 | 0
  Abnormal, NCS, Day 1- 18 hours | 1 | 7
  Abnormal, CS, Day 1- 18 hours | 0 | 0
  Abnormal, NCS, Day 1- 24 hours | 1 | 6
  Abnormal, CS, Day 1- 24 hours | 0 | 0
  Abnormal, NCS, Day 1- 36 hours | 0 | 4
  Abnormal, CS, Day 1- 36 hours | 0 | 0
  Abnormal, NCS, Day 1- 48 hours | 2 | 7
  Abnormal, CS, Day 1- 48 hours | 0 | 0

47. Secondary Outcome: Part 1- Period 1: Total Unchanged Drug (Ae Total) After Single Dose Administration of Gepotidacin 1500 mg
Description: Urine samples were collected at indicated time points for PK analysis. PK parameters were calculated using standard non-compartmental analysis. Ae total was calculated by adding all the fractions of drug collected over all the allotted time intervals.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Milligrams | 328.1 (68.09)

48. Secondary Outcome: Part 1- Period 1: Amount of Drug Excreted in Urine in a Time Interval (Ae[t1-t2]) After Single Dose Administration of Gepotidacin 1500 mg
Description: Urine samples were collected at the specified intervals for PK analysis. PK parameters were calculated using standard non-compartmental analysis. Ae(t1-t2) measured the amount of drug excreted in urine at defined time intervals.
Time Frame: 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Milligrams
  Ae (0-2), n=14 | 50.87 (61.194)
  Ae (2-4), n=13: number analyzed (Participants) | 13
  Ae (2-4), n=13 | 92.98 (51.315)
  Ae (4-6), n=13: number analyzed (Participants) | 13
  Ae (4-6), n=13 | 68.14 (39.927)
  Ae (6-8), n=14 | 47.68 (25.551)
  Ae (8-12), n=14 | 35.71 (11.458)
  Ae (12-24), n=14 | 29.10 (7.8849)
  Ae (24-36), n=13: number analyzed (Participants) | 13
  Ae (24-36), n=13 | 10.72 (4.2330)
  Ae (36-48), n=13: number analyzed (Participants) | 13
  Ae (36-48), n=13 | 5.601 (2.0351)

49. Secondary Outcome: Part 1- Period 1: AUC(0-24) After Single Dose Administration of Gepotidacin 1500 mg (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12 and 12-24 hours post-dose.
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours*micrograms per milliliter | 3340.0 (2340.34)

50. Secondary Outcome: Part 1- Period 1: AUC(0-48) After Single Dose Administration of Gepotidacin 1500 mg (Urine)
Description: Urine samples were be collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours*micrograms per milliliter | 3567.9 (2377.71)

51. Secondary Outcome: Part 1- Period 1: Percentage of the Given Dose of Drug Excreted in Urine (fe%) After Single Dose Administration of Gepotidacin 1500 mg
Description: Urine samples were collected at indicated time points for PK analysis. PK parameters were calculated using standard non-compartmental analysis. fe% was calculated as: (Ae total/Dose) x 100 percent (%).
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Percent dose excreted | 21.874 (4.5393)

52. Secondary Outcome: Part 1- Period 1: Renal Clearance of Drug (CLr) After Single Dose Administration of Gepotidacin 1500 mg
Description: Urine samples were collected at indicated time points for PK analysis. PK parameters were calculated using standard non-compartmental analysis. CLr was calculated as: Ae total/AUC(0-t)
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Liters per hour | 16.66 (3.4123)

53. Secondary Outcome: Part 1- Period 2: Ae Total After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: Urine samples were collected at indicated time points. Ae total were calculated by adding all the fractions of drug collected over all the allotted time intervals.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-14, 14-16, 16-18, 18-20, 20-24, 24-36, 36-48 and 48-60 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Milligrams | 1452.7 (223.10)

54. Secondary Outcome: Part 1- Period 3: Ae Total After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 53
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36, 36-48 and 48-60 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Milligrams | 1293.9 (367.48)

55. Secondary Outcome: Part 1- Period 2: Ae(t1-t2) After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: Urine samples were collected at indicated time points for PK analysis. PK parameters were calculated using standard non-compartmental analysis. Ae(t1-t2) measured the amount of drug excreted in urine at defined time intervals
Time Frame: 0-2, 2-4, 4-6, 6-8, 8-12, 12-14, 14-16, 16-18, 18-20, 20-24, 24-36, 36-48 and 48-60 hours post-dose
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Milligrams
  Ae (0-2), n=13 | 158.5 (81.599)
  Ae (2-4), n=12: number analyzed (Participants) | 12
  Ae (2-4), n=12 | 186.1 (73.777)
  Ae (4-6), n=13 | 143.6 (73.790)
  Ae (6-8), n=12: number analyzed (Participants) | 12
  Ae (6-8), n=12 | 66.80 (22.886)
  Ae (8-12), n=13 | 64.98 (23.987)
  Ae (12-14), n=12: number analyzed (Participants) | 12
  Ae (12-14), n=12 | 204.1 (113.98)
  Ae (14-16), n=13 | 254.3 (83.985)
  Ae (16-18), n=12: number analyzed (Participants) | 12
  Ae (16-18), n=12 | 156.7 (85.023)
  Ae (18-20), n=13 | 80.29 (43.563)
  Ae (20-24), n=13 | 79.23 (25.216)
  Ae (24-36), n=13 | 74.53 (21.862)
  Ae (36-48), n=13 | 20.35 (5.7977)
  Ae (48-60), n=13 | 10.51 (5.0038)

56. Secondary Outcome: Part 1- Period 3: Ae(t1-t2) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 55
Time Frame: 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18 -24, 24-36, 36-48 and 48-60 hours post-dose
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Milligrams
  Ae (0-2), n=12: number analyzed (Participants) | 12
  Ae (0-2), n=12 | 97.51 (70.551)
  Ae (2-4), n=10: number analyzed (Participants) | 10
  Ae (2-4), n=10 | 216.8 (97.543)
  Ae (4-6), n=13 | 172.2 (98.842)
  Ae (6-8), n=12: number analyzed (Participants) | 12
  Ae (6-8), n=12 | 242.3 (138.61)
  Ae (8-10), n=11: number analyzed (Participants) | 11
  Ae (8-10), n=11 | 251.0 (115.23)
  Ae (10-12), n=12: number analyzed (Participants) | 12
  Ae (10-12), n=12 | 151.6 (91.694)
  Ae (12-14), n=12: number analyzed (Participants) | 12
  Ae (12-14), n=12 | 107.3 (77.898)
  Ae (14-18), n=12: number analyzed (Participants) | 12
  Ae (14-18), n=12 | 72.83 (27.363)
  Ae (18-24), n=12: number analyzed (Participants) | 12
  Ae (18-24), n=12 | 63.91 (48.404)
  Ae (24-36), n=13 | 39.13 (12.057)
  Ae (36-48), n=13 | 15.64 (5.9580)
  Ae (48-60), n=13 | 8.889 (4.1747)

57. Secondary Outcome: Part 1- Period 2: AUC(0-tau) (Tau=12 Hours Post-dose) After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8 and 8-12 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 7287.4 (4050.81)

58. Secondary Outcome: Part 1- Period 3: AUC(0-tau) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin
Time Frame: Pre-dose, 0-2, 2-4 and 4-6 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 3943.5 (3015.98)

59. Secondary Outcome: Part 1- Period 2: AUC(0-24) After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-14, 14-16, 16-18, 18-20 and 20-24 hours post dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 17431.6 (10132.84)

60. Secondary Outcome: Part 1- Period 3: AUC(0-24) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18 and 18-24 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 13174.1 (8648.92)

61. Secondary Outcome: Part 1- Period 2: AUC(0-48) After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-14, 14-16, 16-18, 18-20, 20-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 19128.3 (10934.06)

62. Secondary Outcome: Part 1- Period 3: AUC(0-48) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 14277.1 (9045.37)

63. Secondary Outcome: Part 1- Period 2: fe% After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: Urine samples were collected at indicated time points for PK analysis. PK parameters were calculated using standard non-compartmental analysis. fe% was calculated as: (Ae total/Dose) x 100%.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-14, 14-16, 16-18, 18-20, 20-24, 24-36, 36-48 and 48-60 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Percent dose excreted | 24.212 (3.7184)

64. Secondary Outcome: Part 1- Period 3: fe% After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 63
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36, 36-48 and 48-60 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Percent dose excreted | 21.565 (6.1246)

65. Secondary Outcome: Part 1- Period 2: CLr After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: as for outcome 52
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-14, 14-16, 16-18, 18-20, 20-24, 24-36, 36-48 and 48-60 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Liters per hour | 15.88 (2.0305)

66. Secondary Outcome: Part 1- Period 3: CLr After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 52
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36, 36-48 and 48-60 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Liters per hour | 14.81 (3.4456)

67. Secondary Outcome: Part 2- Period 1: Ae Total After Single Dose Administration of Gepotidacin 1500 mg
Description: Urine samples were collected at indicated time points. Ae total was calculated by adding all the fractions of drug collected over all the allotted time intervals
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Milligrams | 361.5 (83.95)

68. Secondary Outcome: Part 2- Period 1: Ae(t1-t2) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 55
Time Frame: 0-2, 2-4, 4-6, 6-8, 8-12, 12-24,24-36 and 36-48 hours post-dose
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Milligrams
  Ae (0-2), n=13 | 16.00 (28.532)
  Ae (2-4), n=12: number analyzed (Participants) | 12
  Ae (2-4), n=12 | 130.5 (49.526)
  Ae (4-6), n=12: number analyzed (Participants) | 12
  Ae (4-6), n=12 | 85.47 (37.814)
  Ae (6-8), n=13 | 58.74 (32.586)
  Ae (8-12), n=13 | 40.15 (14.232)
  Ae (12-24), n=13 | 30.87 (11.638)
  Ae (24-36), n=13 | 10.11 (4.6348)
  Ae (36-48), n=13 | 6.312 (2.5619)

69. Secondary Outcome: Part 2- Period 1: AUC(0-24) After Single Dose Administration of Gepotidacin 1500 mg (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12 and 12-24 hours post-dose.
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 4513.7 (2623.81)

70. Secondary Outcome: Part 2- Period 1: AUC(0-48) After Single Dose Administration of Gepotidacin 1500 mg (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours*micrograms per milliliter | 4948.4 (2721.49)

71. Secondary Outcome: Part 2- Period 1: fe% After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 63
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Percent dose excreted | 24.100 (5.5968)

72. Secondary Outcome: Part 2- Period 1: CLr After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 52
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-12, 12-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Liters per hour | 15.56 (3.7934)

73. Secondary Outcome: Part 2- Period 2: Ae Total After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 67
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Milligrams | 1719.4 (402.71)

74. Secondary Outcome: Part 2- Period 2: Ae(t1-t2) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 55
Time Frame: 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36 and 36-48 hours post-dose
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Milligrams
  Ae (0-2), n=11: number analyzed (Participants) | 11
  Ae (0-2), n=11 | 105.3 (121.67)
  Ae (2-4), n=10: number analyzed (Participants) | 10
  Ae (2-4), n=10 | 202.0 (70.108)
  Ae (4-6), n=10: number analyzed (Participants) | 10
  Ae (4-6), n=10 | 229.7 (113.95)
  Ae (6-8), n=11: number analyzed (Participants) | 11
  Ae (6-8), n=11 | 244.9 (149.66)
  Ae (8-10), n=12 | 446.6 (138.33)
  Ae (10-12), n=10: number analyzed (Participants) | 10
  Ae (10-12), n=10 | 228.3 (79.619)
  Ae (12-14), n=11: number analyzed (Participants) | 11
  Ae (12-14), n=11 | 172.5 (63.150)
  Ae (14-18), n=10: number analyzed (Participants) | 10
  Ae (14-18), n=10 | 132.6 (51.586)
  Ae (18-24), n=10: number analyzed (Participants) | 10
  Ae (18-24), n=10 | 67.56 (40.521)
  Ae (24-36), n=12 | 61.99 (51.367)
  Ae (36-48), n=12 | 14.86 (8.3210)

75. Secondary Outcome: Part 2- Period 2: AUC(0-tau) (Tau=6 Hours Post-dose) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval (Urine)
Description: Urine samples will be collected at indicated time points for pharmacokinetic analysis of gepotidacin
Time Frame: Pre-dose, 0-2, 2-4, 4-6 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter | 5364.4 (2877.94)

76. Secondary Outcome: Part 2- Period 2: AUC(0-24) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin.
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18 and 18-24 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter | 22052.8 (11410.09)

77. Secondary Outcome: Part 2- Period 2: AUC(0-48) After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval (Urine)
Description: Urine samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36 and 36-48 hours post-dose.
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours*micrograms per milliliter | 24500.7 (12281.23)

78. Secondary Outcome: Part 2- Period 2: fe% After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 63
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Percent dose excreted
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Percent dose excreted | 28.657 (6.7119)

79. Secondary Outcome: Part 2- Period 2: CLr After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 52
Time Frame: Pre-dose, 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, 12-14, 14-18, 18-24, 24-36 and 36-48 hours post-dose
Population: PK parameter population
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Liters per hour | 14.93 (3.9558)

80. Secondary Outcome: Part 1- Period 1: Time to Reach Maximum Observed Plasma Concentration (Tmax) After Single Dose Administration of Gepotidacin 1500 mg
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of gepotidacin. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours | 3.000 [0.50 to 6.00]

81. Secondary Outcome: Part 1- Period 1: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours | 0.000 [0.00 to 1.50]

82. Secondary Outcome: Part 1- Period 1: Terminal Phase Half-life (t1/2) After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Gepotidacin 1500 mg
Number analyzed (Participants) | 14
Hours | 11.533 (36.2)

83. Secondary Outcome: Part 1- Period 2: Tmax After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: as for outcome 80
Time Frame: as for outcome 6
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours
  Dose 1 | 2.000 [1.00 to 4.00]
  Dose 2 | 1.567 [1.00 to 4.00]

84. Secondary Outcome: Part 1- Period 3: Tmax After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours
  Dose 1 | 2.633 [0.50 to 5.42]
  Dose 2 | 1.500 [1.00 to 3.28]

85. Secondary Outcome: Part 1- Period 2: Tlag After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: as for outcome 80
Time Frame: as for outcome 6
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours | 0.000 [0.00 to 0.00]

86. Secondary Outcome: Part 1- Period 3: Tlag After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours | 0.000 [0.00 to 0.00]

87. Secondary Outcome: Part 1- Period 2: t1/2 After Two Doses Administration of Gepotidacin 3000 mg at 12 Hour Dosing Interval
Description: as for outcome 80
Time Frame: as for outcome 6
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Gepotidacin 3000 mg 12 Hour Interval
Number analyzed (Participants) | 13
Hours | 10.976 (27.3)

88. Secondary Outcome: Part 1- Period 3: t1/2 After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Dosing Interval
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36, 48 and 60 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 13
Hours | 12.020 (14.6)

89. Secondary Outcome: Part 2- Period 1: Tmax After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours | 3.000 [1.50 to 6.50]

90. Secondary Outcome: Part 2- Period 1: Tlag After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours | 0.500 [0.00 to 1.50]

91. Secondary Outcome: Part 2- Period 1: t1/2 After Single Dose Administration of Gepotidacin 1500 mg
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36 and 48 hours post-dose
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Gepotidacin 1500 mg
Number analyzed (Participants) | 13
Hours | 12.984 (16.6)

92. Secondary Outcome: Part 2- Period 2: Tmax After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours
  Dose 1 | 2.750 [1.00 to 4.00]
  Dose 2 | 1.500 [1.00 to 3.00]

93. Secondary Outcome: Part 2- Period 2: Tlag After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours | 0.000 [0.00 to 0.50]

94. Secondary Outcome: Part 2- Period 2: t1/2 After Two Doses Administration of Gepotidacin 3000 mg at 6 Hour Interval
Description: as for outcome 80
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 6.5, 7, 7.5, 8, 8.5, 9, 10, 12, 14, 18, 24, 36 and 48 hours post-dose
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: Gepotidacin 3000 mg 6 Hour Interval
Number analyzed (Participants) | 12
Hours | 6.982 (19.7)

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from start of study intervention (Day 1) up to Day 19 for Part 1 and up to Day 21 for Part 2.
Description: Safety Population consisted of all participants who received at least 1 dose of study intervention.
Groups:
- Part 1 : Placebo: Adult participants received a single oral dose of gepotidacin matching placebo on Day 1 of Period 1
- Part1: Gepotidacin 1500 mg: Adult participants received a single oral dose of gepotidacin 1500 mg on Day 1 of Period 1
- Part 2 : Placebo: Adolescent participants received a single oral dose of gepotidacin matching placebo on Day 1 of Period 1
Arm/Group | Part 1 : Placebo | Part1: Gepotidacin 1500 mg | Part 1: Gepotidacin 3000 mg 12 Hour Interval | Part 1: Gepotidacin 3000 mg 6 Hour Interval | Part 2 : Placebo | Part 2: Gepotidacin 1500 mg | Part 2: Gepotidacin 3000 mg 6 Hour Interval
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/14 | 0/13 | 0/13 | 0/3 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/14 | 0/13 | 0/13 | 0/3 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/2 | 1/14 | 10/13 | 9/13 | 2/3 | 9/14 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 : Placebo (N=2) | Part1: Gepotidacin 1500 mg (N=14) | Part 1: Gepotidacin 3000 mg 12 Hour Interval (N=13) | Part 1: Gepotidacin 3000 mg 6 Hour Interval (N=13) | Part 2 : Placebo (N=3) | Part 2: Gepotidacin 1500 mg (N=14) | Part 2: Gepotidacin 3000 mg 6 Hour Interval (N=12)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 8 (8) | 8 (8) | 1 (1) | 3 (3) | 5 (5)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 1 (2) | 0 (0) | 9 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT04079790/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT04079790/SAP_001.pdf